CLINICAL TRIAL: NCT03647462
Title: The Impact of Early Diagnosis and Treatment of OSA on Hospital Readmission in Hospitalized Chronic Obstructive Pulmonary Disease Patients: the COPD Readmit Clinical Trial
Brief Title: Impact of Early Diagnosis and Treatment of OSA on Hospital Readmission in Hospitalized COPD Patients
Acronym: COPD Readmit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Dennis Hwang, MD, Medical Director, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPSleep-004
Record Dates: First submitted 2018-08-08; First posted 2018-08-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease
Keywords: obstructive sleep apnea; chronic obstructive sleep apnea; hospital readmission
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPAP Intervention Pathway (Experimental): Patients will receive continuous positive airway pressure (CPAP) therapy in the hospital followed by home CPAP therapy. Their home CPAP therapy will include wireless connectivity, which includes adherence data. Furthermore, the patients will be entered into our usual automated platform (USleep; ResMed Corp) in which patients with suboptimal CPAP use will be sent messages (based on patient preference) in order to ensure adherence to therapy. This platform is already a standard part of our usual care.
  The patients will receive CPAP in addition to contemporary standard of care pharmacotherapy for their underlying COPD. They will follow up at the Fontana Sleep Center within 1 month after discharge for assessment of CPAP use and asked to complete a questionnaire packet. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms.
  Interventions: Device: Continuous Positive Airway Pressure
- Usual Care Pathway (No Intervention): Patients will receive contemporary standard of care pharmacotherapy for their underlying COPD condition and will not receive CPAP therapy for the duration of the study. They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for a repeat outpatient portable sleep study and asked to complete a questionnaire packet. The results of the outpatient portable sleep studies will be compared with the in-patient portable sleep study. Patients will also be asked to follow up with the Fontana Sleep Center within 1 month after discharge for assessment of primary and secondary outcomes. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP is an FDA approved therapy machine for patients diagnosed with OSA. CPAP provides positive air pressure to the patients throat to ensure the patients airway stays open during sleep. CPAP is the gold standard treatment for OSA, but there is limited research that demonstrates whether CPAP can improve clinical outcomes in patients with COPD. Therefore, our investigators want to initiate CPAP therapy in patients hospitalized for COPD to investigate whether there is an improvement in cardiac function and clinical outcomes (i.e. mortality).
  Other Names: CPAP; APAP
  Arms: CPAP Intervention Pathway

SUMMARY:
The purpose of this study is to determine whether early diagnosis of OSA and initiation of and adherence to CPAP therapy in patients hospitalized for chronic obstructive pulmonary disease reduce 30-day hospital readmission rates.

DETAILED DESCRIPTION:
Our investigators propose a randomized clinical trial to test hospitalized patients (due to chronic obstructive pulmonary disease, COPD) for obstructive sleep apnea, then randomizing the patients with OSA into CPAP versus usual care. This study is designed to target a high risk population (hospitalized patients) and early initiation of therapy. Our investigators intend to enroll all consenting participants hospitalized with a primary COPD diagnosis. Our study is unique and the answer to its question - whether early diagnosis of OSA and initiation of and adherence to CPAP therapy in hospitalized COPD patients will reduce 30-day readmission rates - is unknown. The objective is twofold: to improve quality of care and decrease preventable hospitalizations through early diagnosis and implementation of this early diagnosis and intervention model for this subset of patients may slow progression of COPD, offset a large public health and financial burden, and improve overall outcomes.

Our investigators believe that our study, which involves human subjects, is in accordance with general ethical principles. It should be noted that the diagnosis and subsequent treatment of OSA during hospitalization is not part of routine practice, and that the control group truly would follow "usual care". Moreover, patients who are deemed very sick (as outlined in the exclusion criteria) will be excluded from the study. Finally half of enrolled participants will receive early CPAP therapy which may potentially benefit those patients beyond what is currently "usual care".

Study Design

Our study is a single-center, randomized control trial designed to evaluate the impact of early diagnosis and treatment of obstructive sleep apnea (OSA) in hospitalized chronic obstructive pulmonary disease (COPD) patients on hospital readmission, symptoms, and healthcare utilization. Consecutive patients who meet inclusion criteria hospitalized with a primary diagnosis of COPD will be asked to participate in the study. Patients who agree and sign consent will undergo a portable sleep study to diagnose OSA-predominant sleep disordered breathing. Patients will also complete a questionnaire packet consisting of the following standardized questionnaires: sleep history questionnaire, Epworth Sleepiness Scale (ESS), Patient Recorded Outcome Measurement Information System (PROMIS), Chronic Obstructive Pulmonary Disease Assessment Tool (CAT), and STOP-BANG questionnaire. Each patient who meets inclusion criteria and consents to the study will undergo an inpatient portable sleep study (ApneaLink, Resmed Corp). This is a Type III study which is an unattended study that measures nasal pressure, respiratory effort, oxygen saturation, and body position. A study investigator will apply the portable device, and a board-certified sleep medicine physician (co-investigators) will interpret these studies. The study will be performed while the patient is on room air (not on oxygen), thus the study may not be applied on the first hospitalized night (if oxygen therapy is required) but delayed until the patient is appropriate to be off oxygen.

A diagnosis of OSA will be made if the apnea-hypopnea index with 4% oxygen desaturation is greater than 5 (AHI4%≥5) with at least 50% of events consistent with obstructive rather than central physiology. Study participants with OSA will then be randomized into one of two pathways: Intervention Pathway and Usual Care Pathway.

Intervention Pathway Patients will receive CPAP therapy in the hospital followed by home CPAP therapy. A sleep center respiratory therapy/sleep technologist case manager will perform a bedside mask fit, CPAP education, and set up their outpatient follow-up appointments with the sleep center. Their home CPAP therapy will be a loaner from the sleep medicine department that includes wireless connectivity so that adherence data is available to the investigators throughout the duration of the study. Furthermore, the patients will be entered into our usual automated platform (USleep; ResMed Corp) in which patients with suboptimal CPAP use will be sent messages (email or text based on patient preference) in order to ensure adherence to therapy. This platform is already a standard part of our usual care.

The patients will receive CPAP in addition to the contemporary standard of care pharmacotherapy for their underlying cardiac condition(s). They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for assessment of CPAP use and asked to complete the aforementioned questionnaire packet (with the exception of the STOP BANG questionnaire). Patients will also be asked to follow up within 30 days after discharge for assessment of CPAP use and asked to complete the aforementioned questionnaire packet. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms. During the 1 month follow-up appointment, the sleep center will troubleshoot CPAP use when appropriate; otherwise, requests for additional troubleshooting will be at the discretion of the patient (as is currently our usual care).

Usual Care Pathway Patients will receive contemporary standard of care pharmacotherapy for their underlying cardiac condition(s) and will not receive CPAP therapy for the duration of the study. They will be asked to follow up at the Fontana Sleep Center within 1 month after discharge for a repeat outpatient portable sleep study and asked to complete the aforementioned questionnaire packet (with the exception of the STOP BANG questionnaire). The results of the outpatient portable sleep studies will be compared with the in-patient portable sleep study. Patients will also be asked to follow up with the Fontana Sleep Center within 30 days after discharge for assessment of primary and secondary outcomes. Patients will be followed during the 30-day period and assessed for readmission rates, time to readmission, adherence to CPAP therapy, and presence of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente member
* Males or females, any race, and age 18 and older
* OSA-predominant (AHI at or above 5) sleep disordered breathing
* Primary diagnosis upon admission of chronic obstructive pulmonary disease
* Appropriate to perform portable sleep study while on room air (no oxygen)
* Patients who are able and willing to give informed consent

Exclusion Criteria:

* Use of CPAP within 6 months of enrollment
* Patients with CSA-predominant sleep disordered breathing
* Patients who are "sleepy": ESS at or above 11
* Commercial driver's license or other occupational hazards (operating heavy machinery)
* Non-English speaking (validated questionnaires are currently limited to English)
* Patients with chronic respiratory failure requiring oxygen therapy or non-invasive ventilation.
* Patients requiring tracheostomy
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Hospital readmission and mortality rates | 30 days
  Number of occasions patient has been admitted to the hospital and number of patients who have died

SECONDARY OUTCOMES:
Clinic and urgent care visits | 30 days
  Appointments with any medical providers (sleep, cardiac, primary) at a clinic or urgent care facility
Off work orders | 30 days
  Note from provider ordering/requesting patient to be dismissed from work for medical reasons (sick, injured, etc.)
STOP BANG | 30 days
  Snoring, tiredness, observed apnea, blood pressure, body mass index, age, neck circumference, and gender (STOP BANG) is the name of a OSA screening questionnaire. Questionnaire contains 8 "Yes/No" questions and the number of "Yes" answers provide a total score (range 0-8). Patients that answer "Yes" to 3-4 questions are typically considered to be at intermediate risk of OSA.
Epworth Sleepiness Scale (ESS) | 30 days
  Epworth Sleepiness Scale measures degree of sleepiness. 8 scenarios are described and the responder indicates their likelihood of dozing unintentionally (range 0-3). A total of the scores are added (range 0-24) and typically scores of at least 11 indicate excessive sleepiness.
Patient Reported Outcome Measurement Information System (PROMIS) | 30 days
  Patient Reported Outcome Measurement Information System is a 10 item questionnaire that measures physical, mental, and social health in adults. It can be used on the general population and patients with chronic conditions. Patients rate their health based on a severity scale of 1-5 (1 indicates poor health) and the scoring system allows each question/item to be evaluated separately.
Chronic Obstructive Pulmonary Disease Assessment Tool (CAT) | 30 days
  Chronic Obstructive Pulmonary Disease (COPD) Assessment Tool is a questionnaire that measures the impact the disease has on patients well being and daily life. There are 8 questions that ask about common symptoms COPD patients experience and the patient indicates their severity (range 0-5). A total of the scores are added (range 0-40) and scores of at least 30 indicate that their COPD has a very high level of impact on their daily lives.
Comparing inpatient portable monitor versus 30-day follow up portable monitor results in usual care group | 30 days
  Evaluating the change of sleep diagnostic test results from the hospital to 1-month after being discharged (only for patients enrolled in the Usual Care pathway)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente, Fontana Medical Center
Locations (1):
- Sleep Center; San Bernardino County Medical Center, Kaiser Permanente, Fontana, California, United States